CLINICAL TRIAL: NCT01824056
Title: The Differential Diagnosis of Parkinson's Disease and Parkinsonism by Positron-emission Tomography With Vesicular Monoamine Transporter Ligand (18F-DTBZ)
Brief Title: The Differential Diagnosis of Parkinson's Disease and Parkinsonism by Positron-emission Tomography
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, NJI90OKM, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 98-3626A
Record Dates: First submitted 2013-03-12; First posted 2013-04-04 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson's Disease
Keywords: 18F-FDG
MeSH Terms: conditions — Parkinson Disease | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DTBZ for Parkinson's Disease (Experimental): This study will compare the brain uptake of 18F- DTBZ in 40 patients with PD, 40 patients with MSA, 20 patients with CBD, and 20 patients with PSP . Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, each subject will have 3 visits in this study. Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — During this study, subjects will receive a single i.v. administration of approximately 10 mCi 18F-FP-(+)-DTBZ immediately prior to imaging.
  The proposed dose for this study is based on our phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG.

SUMMARY:
The objective of this protocol is to analyze the sensitivity and specificity of 18F-DTBZ PET to the differential diagnosis of Parkinson's disease (PD) and other parkinsonism disorders, including multiple system atrophy (MSA), corticobasal degeneration (CBD), and progressive supranuclear palsy (PSP).

DETAILED DESCRIPTION:
40 patients with PD, 40 patients with MSA, 20 patients with CBD, and 20 patients with PSP, will be enrolled. Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, each subject will have 3 visits in this study, as one screening visit, one imaging visit, and one safety evaluation visit.

Safety measurement will be evaluated by medical history, vital signs, physical examinations,

ELIGIBILITY:
Inclusion Criteria:

1. Forty subjects with a diagnosis of PD whom must:

   i.Male or female patients, age range 20~80. ii.Patients should be fulfilled Criteria of diagnosis of Parkinson disease8 of "possible" or "probable" PD (Appendix I).

   iii.Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
2. Forty subjects with a diagnosis of MSA whom must:

   i.Male or female patients, age range 20~80. ii.Patients should be fulfilled the Consensus diagnostic criteria of "possible" or "probable" MSA14 (Appendix II).

   iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
3. Twenty subjects with a diagnosis of PSP whom must:

   i.Male or female patients, age range 20~80. ii.Patients should be fulfilled the NINDS-SPSP clinical criteria for the diagnosis of PSP of "possible" or "probable" PSP35 (Appendix III).

   iii.Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).
4. Twenty subjects with a diagnosis of CBD whom must:

   i.Male or female patients, age range 20~80. ii.Patients should be fulfilled the Kumar's criteria of CBD36 (Appendix IV). iii.Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study or current breast feeding.
2. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.

   i.Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances.

   ii.Current clinically significant cardiovascular disease. (cardiac surgery or myocardial infarction within the last 6 months; unstable angina; decompensated congestive heart failure; significant cardiac arrhythmia; congenital heart disease.
3. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
4. History or presence of QTc prolongation.
5. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
6. Any documented abnormality in the brain by CT or MRI of brain, which might contribute to the motor function, such as hydrocephalus, multiple infarction and encephalomalacia, will be excluded. Mild cortical atrophy and non-specific white matter changes will be allowed.
7. Patients who have the evidence of secondary parkinsonism (multiple infarcts, intoxication, and hydrocephalus, etc) or other neurodegenerative diseases, such as spinocerebellar atrophy (SCA), Wilson's disease, hydrocephalus, multiple infarction, serious head injury and definite history of neurotoxin exposure, are excluded.
8. General PET exclusion criteria.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To analyze the sensitivity and specificity of 18F-DTBZ PET to the differential diagnosis of PD ,PSP,MSA,CBD. | 3 years
  All subjects that received 18F-FP-(+)-DTBZ for injection.Sensitivity and specificity analysis of VMAT2 imaging will include all subjects for whom there is sufficient data to evaluate the parameter in question.Descriptive statistics will be presented to help detect changes within groups or differences between groups (PD vs. MSA, CBD, PSP). The descriptive statistics will include mean, standard deviation, median, and ranges for continuous variables, and frequency and percent frequency for categorical variables.Mann Whitney test will be used to compare the mean SUVR values between PD and other groups. ROC curve will be used to determinate the diagnostic threshold of SUVR and the sensitivity and specificity of 18F- DTBZ PET in the differentiating PD, MSA, PSP, and CBD. Statistical analysis was performed using a unpaired t test based on one contrast to test a hypothesis of regional abnormal uptakes of 18F-DTBZ in an individual MSA/PSP/CBD patient compared to a PD group.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memory Hpspital, Taoyuan District, Taiwan, Taiwan